CLINICAL TRIAL: NCT07112248
Title: A Randomized Controlled Trial Investigating the Effects of Soluble Dietary Fiber Supplements on Sperm Quality Parameters in Males With Obesity
Brief Title: Effects of Soluble Fiber Supplements on Sperm Quality in Males With Obesity: a Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, PhD, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XXM2025157
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Obesity-related Poor Sperm Quality; Gut Microbiota
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): 1.5 g maltodextrin in a sachet once daily for 12 weeks.
  Interventions: Dietary Supplement: Placebo
- Soluble dietary fiber group (Experimental): 1.5 g inulin in a sachet once daily for 12 weeks.
  Interventions: Dietary Supplement: inulin

INTERVENTIONS:
Dietary Supplement: Placebo — Maltodextrin
  Arms: Control group
Dietary Supplement: inulin — Inulin is a kind of soluble dietary fiber.
  Arms: Soluble dietary fiber group

SUMMARY:
Obesity-related poor sperm quality is a significant public health issue, acting as a major contributor to male infertility. Dietary intervention has emerged as an effective strategy to manage obesity and improve sperm quality. Soluble dietary fiber (SDF), an essential nutritional component, plays a crucial role in regulating host health. Notably, insufficient SDF intake has been associated with both obesity and low sperm motility. However, the effect of SDF supplementation on sperm quality in males with obesity remains unclear. Thus, we conducted a randomized, placebo-controlled study to investigate the effect of SDF supplementation on sperm quality in males with obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged 18-60 years；
2. Diagnostic criteria for obesity: BMI ≥ 28 kg/m² and body fat percentage ≥ 25%;
3. Semen samples can be collected, and sperm concentration > 0.

Exclusion Criteria:

1. Spermatogenic dysfunction caused by non-obesity factors;
2. Severe systemic diseases such as cardiovascular/cerebrovascular, hepatic/renal disorders, malignant tumors, uncontrolled diabetes, or thyroid diseases;
3. Recent usage of medications/supplements affecting spermatogenesis or gut microbiota ;
4. Lifestyle factors potentially impairing sperm quality or severe gastrointestinal disorders;
5. Poor compliance, planned imminent fertility, or history of bariatric surgery/weight-loss medications;
6. Significant dietary changes within the past three months.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The sperm quality of obese males | Baseline, 4 weeks and 12 weeks.
  The sperm quality includes the motility, concentration and morphology of sperm and these parameters are all measured by Computer-Assisted Semen Analysis.

SECONDARY OUTCOMES:
Changes in the levels of sex hormones | Baseline, 4 weeks, 12 weeks
  Changes in the levels of sex hormones, including Follicle-Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2), Progesterone (P), Testosterone (T), and Prolactin (PRL).
Changes in sexual function | Baseline, 4 weeks, 12 weeks
  The sexual function will be assessed by Brief Male Sexual Function Questionnaire.
Changes in DNA integrity of sperm | Baseline, 4 weeks, 12 weeks
  Changes in the sperm DNA fragmentation index (DFI) will be measured by sperm chromatin structure assay (SCSA).
Changes in the gut microbiota | Baseline, 4 weeks, 12 weeks
  Changes in the composition, diversity, and function of gut microbiota in feces will be measured by 16S rRNA gene sequencing.
Changes in the levels of bile acids in plasma | Baseline, 4 weeks, 12 weeks
  Changes in the levels of bile acids in plasma will be evaluated by liquid chromatography-mass spectrometry (LC-MS).
Changes in the levels of fasting plasma TC, TG, LDL, and HDL | Baseline, 4 weeks, 12 weeks
Change in body weight | Baseline, 4 weeks, 12 weeks
Change in BMI | Baseline, 4 weeks, 12 weeks
Change in waist-to-hip ratio (WHR) | Baseline, 4 weeks, 12 weeks
Change in body fat composition | Baseline, 4 weeks, 12 weeks
Change in the levels fasting plasma glucose | Baseline, 4 weeks, 12 weeks